CLINICAL TRIAL: NCT07331142
Title: Efficacy and Safety of Prophylactic Biliary Stenting After Complete Common Bile Duct Stone Clearance Before Cholecystectomy: A Randomized Controlled Trial
Brief Title: CBD Stenting vs Non-Stenting for Choledocholithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 035931299
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Choledocholithiasis
Keywords: Choledocholithiasis; cholelithiasis; endoscopic retrograde cholangiopancreatography; stent
MeSH Terms: conditions — Choledocholithiasis; Cholelithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic Biliary Stenting Group (Experimental): Patients randomized to this arm receive endoscopic placement of a temporary plastic biliary stent (7-10 French) in the common bile duct after documented complete choledocholithiasis clearance during ERCP. The stent is left in place to maintain bile duct patency during the waiting period before cholecystectomy.
  Interventions: Procedure: Temporary Plastic Biliary Stent Placement; Procedure: Endoscopic Retrograde Cholangiopancreatography with Stone Clearance
- No Stenting Group (Active Comparator): Patients randomized to this arm undergo ERCP with complete choledocholithiasis clearance without placement of a temporary biliary stent. They proceed to laparoscopic cholecystectomy without the protective stent.
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography with Stone Clearance

INTERVENTIONS:
Procedure: Temporary Plastic Biliary Stent Placement — Endoscopic placement of a temporary plastic biliary stent (7-10 French gauge) across the sphincter of Oddi after documented complete choledocholithiasis clearance on occlusion cholangiogram during ERCP. The stent maintains bile duct patency and is left in place until cholecystectomy.
  Arms: Prophylactic Biliary Stenting Group
Procedure: Endoscopic Retrograde Cholangiopancreatography with Stone Clearance — Standard endoscopic retrograde cholangiopancreatography (ERCP) with endoscopic sphincterotomy and complete choledocholithiasis clearance documented on occlusion cholangiogram. No temporary biliary stent is placed.

SUMMARY:
The role of prophylactic biliary stenting after complete clearance of common bile duct stones in patients awaiting cholecystectomy remains controversial. This randomized controlled trial investigates whether temporary plastic biliary stent placement after documented complete choledocholithiasis clearance reduces the recurrence of choledocholithiasis and biliary complications in patients awaiting cholecystectomy for concomitant cholelithiasis.

Between March 2024 and September 2025, 200 patients with concomitant cholelithiasis and choledocholithiasis were randomized to either prophylactic biliary stenting (n=100) or no stenting (n=100) after complete stone clearance documented on occlusion cholangiogram during endoscopic retrograde cholangiopancreatography (ERCP).

The primary outcome was symptomatic choledocholithiasis recurrence within 3 months. Secondary outcomes included biliary complications (cholangitis, cholecystitis, post-ERCP pancreatitis, bleeding), radiation exposure metrics, and cost-effectiveness.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Choledocholithiasis frequently coexists with cholelithiasis and is typically managed through a two-stage approach: endoscopic retrograde cholangiopancreatography (ERCP) for stone clearance, followed by laparoscopic cholecystectomy to remove the source of stone formation. The timing and sequencing of these procedures, as well as the role of temporary protective measures during the interval between ERCP and cholecystectomy, have been subjects of clinical debate.

Prophylactic biliary stenting after complete stone clearance has been suggested as a potential protective measure to maintain bile duct patency and prevent recurrent stone migration during the waiting period before cholecystectomy. The theoretical advantages include prevention of stent-related complications such as post-ERCP pancreatitis, maintenance of adequate bile drainage, and reduction in recurrent biliary events. However, the actual clinical benefit of this practice has not been definitively established, and temporary stents themselves carry risks including stent occlusion, migration, and infection.

STUDY OBJECTIVES:

Primary Objective: To determine whether prophylactic biliary stent placement after documented complete choledocholithiasis clearance reduces the recurrence of choledocholithiasis in patients awaiting cholecystectomy.

Secondary Objectives: To compare the incidence of biliary complications (cholecystitis, post-ERCP pancreatitis, cholangitis) between the stenting and no-stenting groups, to assess the need for repeat or emergency ERCP during the follow-up period, to evaluate stent-related complications in the stenting group, and to compare radiation exposure metrics, and cost-effectiveness.

STUDY DESIGN:

This is a prospective, randomized controlled trial with parallel assignment comparing prophylactic biliary stenting versus no stenting in patients with complete choledocholithiasis clearance awaiting cholecystectomy. The study is open-label, with outcome assessors blinded to treatment allocation.

STUDY POPULATION:

The study includes adult patients (age 18-75 years) with concomitant cholelithiasis and choledocholithiasis who have undergone successful ERCP with complete stone clearance documented on occlusion cholangiogram. Patients are excluded if they have incomplete stone clearance, altered anatomy precluding stent placement, active cholangitis, immunocompromised status, or contraindications to cholecystectomy.

RANDOMIZATION AND ALLOCATION:

Participants are randomized 1:1 to either the stenting group or the no-stenting group using a computer-generated randomization sequence with permuted blocks. Randomization is stratified by study site to ensure balanced allocation across participating centers. Allocation concealment is maintained through sealed, opaque envelopes.

INTERVENTIONS:

Stenting Group: Following successful ERCP with complete choledocholithiasis clearance (documented on occlusion cholangiogram), a temporary plastic biliary stent (7-10 French) is placed across the sphincter of Oddi to maintain bile duct patency until cholecystectomy.

No-Stenting Group: Patients undergo ERCP with complete choledocholithiasis clearance without placement of a temporary biliary stent and proceed directly to cholecystectomy.

FOLLOW-UP PROCEDURES:

All participants are scheduled for laparoscopic cholecystectomy within 2-4 weeks of ERCP. Clinical assessments are performed at baseline (ERCP), week 1, pre-cholecystectomy (week 2-4), and at 1 month and 3 months post-ERCP. Imaging studies (ultrasound or CT) are performed at baseline and at the 3-month follow-up to assess for stone recurrence.

OUTCOME MEASURES:

Primary Outcome: Recurrence of choledocholithiasis documented on imaging or endoscopy during the 3-month follow-up period.

Secondary Outcomes: Incidence of biliary complications (cholecystitis, post-ERCP pancreatitis, cholangitis); need for repeat or emergency ERCP; stent-related complications; hospital readmission rates; time to cholecystectomy.

STATISTICAL ANALYSIS:

The primary analysis compares the recurrence rate between the two groups using chi-square test or Fisher's exact test. Secondary outcomes are compared using appropriate statistical tests. Intention-to-treat analysis is performed, including all randomized participants in their assigned groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years at the time of enrollment
2. Diagnosis of concomitant cholelithiasis and choledocholithiasis
3. Successful ERCP with complete choledocholithiasis clearance documented on occlusion cholangiogram during the index procedure
4. Endoscopic sphincterotomy (EST) performed during ERCP
5. Ability to provide informed consent
6. Scheduled for laparoscopic cholecystectomy within 2-4 weeks of ERCP
7. No contraindications to cholecystectomy

Exclusion Criteria:

1. Incomplete choledocholithiasis clearance (residual stones on occlusion cholangiogram)
2. Altered biliary anatomy (e.g., previous bilioenteric anastomosis, Roux-en-Y reconstruction)
3. Active cholangitis or sepsis at the time of ERCP
4. Immunocompromised status (HIV/AIDS, active chemotherapy, chronic corticosteroid use)
5. Coagulopathy or anticoagulation therapy that cannot be safely interrupted
6. Pregnancy or lactation
7. Severe cardiopulmonary disease precluding safe anesthesia
8. Contraindications to cholecystectomy (e.g., unresectable malignancy, severe cirrhosis with portal hypertension)
9. Participation in another clinical trial within the past 30 days
10. Unable or unwilling to comply with follow-up protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of Choledocholithiasis | 3 months after initial ERCP
  Radiological or endoscopic evidence of recurrent common bile duct stones documented on imaging (ultrasound, CT, MRCP) or during repeat endoscopy.

SECONDARY OUTCOMES:
Biliary Complications | 3 months after initial ERCP
  Incidence of post-ERCP pancreatitis, cholecystitis, cholangitis, or other biliary-related adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Menoufia University, Egypt., Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhu J, Li G, Du P, Zhou X, Xiao W, Li Y. Laparoscopic common bile duct exploration versus intraoperative endoscopic retrograde cholangiopancreatography in patients with gallbladder and common bile duct stones: a meta-analysis. Surg Endosc. 2021 Mar;35(3):997-1005. doi: 10.1007/s00464-020-08052-y. Epub 2020 Oct 6. PMID 33025251
- [Background] Chaudhary S. Epidemiology of gall stone diseases among patients attending surgical department of a tertiary care hospital in Nepal. Janaki Med. Coll. J.Med. Sci., 2020; 8(1), 50-55.
- [Background] Cai H, Sun D, Sun Y, Bai J, Zhao H, Miao Y. Primary closure following laparoscopic common bile duct exploration combined with intraoperative cholangiography and choledochoscopy. World J Surg. 2012 Jan;36(1):164-70. doi: 10.1007/s00268-011-1346-6. PMID 22086256
- [Background] Abd El Wahab AE, Khalil OO. Comparative study between primary common bile duct repair with internal stent insertion versus t-tube drainage after common bile duct exploration. Al-Azhar Intern. Med. J., 2022; 3(1), 107-111.